CLINICAL TRIAL: NCT07143955
Title: A Randomized Controlled Trial of a Targeted Dietary Intervention to Reshape Gut Microbiota and Lipid Metabolism for Enhancing Anti-Tumor Immunity and Prognosis in Patients With Hepatocellular Carcinoma
Brief Title: Dietary Intervention and Gut Microbiota in Hepatocellular Carcinoma (HCC)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Hospital of Hebei Medical University (Other)
Responsible Party: Principal Investigator, Feifei Wang, Principal investigator, The First Hospital of Hebei Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022S00117
Record Dates: First submitted 2025-08-13; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Hepatocellular Carcinoma (HCC)
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Targeted Dietary Intervention Group (Experimental): Patients received routine care plus a structured dietary intervention for the duration of follow-up. The intervention included: 1) A diet plan emphasizing high-fiber foods and lean proteins; 2) A daily multi-species probiotic supplement (≥1x10¹⁰ CFU/day); 3) Encouraged intake of prebiotics (inulin, fructooligosaccharides) and unsaturated fatty acids.
  Interventions: Behavioral: Structured Dietary Intervention
- Active Comparator: Control Group (Active Comparator): Patients received routine dietary care and counseling according to institutional guidelines for HCC patients. This included general advice on maintaining adequate caloric and protein intake.
  Interventions: Behavioral: Routine Dietary Care

INTERVENTIONS:
Behavioral: Structured Dietary Intervention — A comprehensive dietary program consisting of dietary modification (high-fiber, lean protein), daily probiotic supplementation capsule (Bifidobacterium longum, Lactobacillus acidophilus, and Lactobacillus rhamnosus), and encouraged intake of prebiotics and unsaturated fatty acids.
  Arms: Experimental: Targeted Dietary Intervention Group
Behavioral: Routine Dietary Care — Standard institutional dietary counseling for patients with HCC, providing general advice on nutrition.
  Arms: Active Comparator: Control Group

SUMMARY:
This prospective, randomized controlled trial investigates the efficacy of a targeted dietary intervention in patients with hepatocellular carcinoma (HCC). The study aims to compare a structured diet including probiotics and prebiotics against routine dietary care. The primary goal is to assess the impact on clinical outcomes (survival), gut microbiota composition, systemic lipid metabolism, and anti-tumor immune responses, to determine if this intervention can serve as an effective adjunctive therapy for HCC.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is associated with gut microbiota dysbiosis, which contributes to a pro-inflammatory and immunosuppressive tumor microenvironment via the "gut-liver axis." This study hypothesizes that modulating the gut microbiota through a targeted dietary intervention can rebalance systemic immunity and improve clinical outcomes. This single-center, prospective trial randomized 100 patients with HCC into two groups. The experimental group (n=50) received a structured dietary plan including high-fiber foods, probiotics (Bifidobacterium, Lactobacillus), and prebiotics. The control group (n=50) received routine dietary counseling. The study evaluates the intervention's effects on progression-free survival (PFS), overall survival (OS), gut microbiota diversity, serum lipid profiles, peripheral immune cell populations (CD8+ T cells, Tregs), and quality of life. The findings aim to provide robust clinical evidence for integrating microbiota-targeted dietary therapy into the standard management of HCC.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years.
* Pathologically confirmed primary Hepatocellular Carcinoma (HCC).
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
* Adequate organ function (e.g., liver, renal, and bone marrow).
* Life expectancy of at least 3 months.
* Willingness to provide informed consent and adhere to study procedures.

Exclusion Criteria:

* Concurrent malignancies other than HCC.
* Severe, uncontrolled comorbidities (e.g., congestive heart failure, renal failure).
* Known history of severe intestinal diseases such as inflammatory bowel disease.
* Use of antibiotics, probiotics, or other microbiota-altering agents within 4 weeks prior to enrollment.
* Cognitive impairment precluding understanding of the study.
* Refusal to provide consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | Through study completion, an average of 12 months
  Defined as the time from randomization to the first documented disease progression or death from any cause, whichever occurred first. Disease progression was assessed according to standard oncologic criteria.
Overall Survival (OS) | Through study completion, an average of 12 months
  Defined as the time from randomization to death from any cause.

SECONDARY OUTCOMES:
Change in Gut Microbiota Alpha-Diversity | Baseline, 12 months
  Measured by the Shannon and Simpson indices from fecal samples using 16S rRNA sequencing.
Change in Gut Microbiota Composition | Baseline, 12 months
  Relative abundance of key bacterial genera (e.g., Bifidobacterium, Lactobacillus, Escherichia coli) assessed by 16S rRNA sequencing.
Change in Serum Lipid Profile | Baseline, 12 months
  Measured levels of serum cholesterol and triglycerides.
Change in Health-Related Quality of Life (QOL) | Baseline, 12 months
  Assessed using the World Health Organization Quality of Life (WHOQOL-100) questionnaire. Scores for each domain range from 4 to 20, with higher scores indicating a better quality of life.
Incidence of Treatment-Related Adverse Events | Throughout the study duration, up to 18 months
  Safety and tolerability assessed by documenting adverse events throughout the study.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Hebei Medical University, Shijiazhuang, Hebei, China